CLINICAL TRIAL: NCT06887816
Title: Clinical Investigation of the Efficacy of New Silver-coated Prosthesis in Reducing the Incidence of Periprosthetic Infections
Brief Title: Efficacy of New Silver-coated Prosthesis in Reducing the Incidence of Periprosthetic Infections
Status: Recruiting | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Other Study IDs: Silver ProTect
Record Dates: First submitted 2025-03-10; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Hip Infection
Keywords: silver coating; primary prosthesis; second stage surgery

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood draw and urine sample will be collected at the baseline and at the follow-ups (6, 12 and 24 months) for the quantification of silver content with ICP-MS analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Revision patients with outcomes of previous infection awaiting access to "second-stage" surgery or patients awaiting primary prosthetic surgery with recurrent urinary, pulmonary or other district infections.
  Interventions: Device: silver coated device; Device: not silver coated device

INTERVENTIONS:
Device: silver coated device — Patients who will be implanted with prosthesis with a silver coating to counteract infection relapse
Device: not silver coated device — Patients who will be implanted with prosthesis without silver coating

SUMMARY:
The aim of the present clinical study, of prospective observational nature with biological study, is to conduct a clinical investigation on the the efficacy of a device coated with bacteriostatic silver coating, with the overall objective of understand whether the device is indeed able to reduce the number of peri-operative and post-operative infections, both early and late.

DETAILED DESCRIPTION:
Among the various complications that can arise in orthopaedics following implant surgery, peri-prosthetic joint infections (Periprosthetic Joint Infection -PJI) represent one of the most feared complications and the main cause of revision surgeries (15% and 25% of hip and knee revision surgeries, respectively). In this complex context, prevention therefore plays a fundamental role and is a key objective considering the increasing number of patients considered to be at high risk such as the elderly, patients with recurrent infections (urinary, pulmonary, etc.), those suffering from diabetes mellitus or obese, the immunocompromised, or patients who have already undergone prosthetic surgery.

In order to reduce the risk of infection, it is therefore essential to adopt and implement preventive strategies that also involve the medical devices themselves, such as the development of passive surfaces capable of counteracting bacterial adhesion or active surfaces capable of exerting a direct action on micro-organisms. To achieve this second type of action, antibacterial agents, such as silver, known for its antimicrobial and bactericidal properties, are used.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years;
* Immunocompromised patients and/or diabetic patients.
* Patients who have given consent

Exclusion Criteria:

* Patients aged < 18 years;
* Pregnant women;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Revision patients with a history of previous infection awaiting access to 'second-stage' surgery or patients awaiting primary prosthetic surgery with recurrent urinary, pulmonary or other infections will be enrolled
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-03-12 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Number of infections | at 1 month follow-up, at 3 months follow-up, at 6 months follow-up, at 12 months follow-up, at 24 months follow-up
  To evaluate the performance of the silver-coated device in reducing the incidence of early (occurring within 30 days of surgery) and late (occurring more than 90 days after surgery) infectious event in patients considered to be at high risk because they are awaiting primary prosthetic surgery but i) subject to recurrent occurrence of urinary pulmonary or other tract infections, (ii) immunocompromised, (iii) with rheumatic diseases, (iv) diabetics, or spacer carriers awaiting second-stage surgery for previous prosthetic revision due to infection.
Safety profile of silver | day 0 (at baseline), at 6 months follow-up, at 12 months follow-up, at 24 months follow-up
  To assess the safety profile of device prosthesis system in terms of silver release. Blood sampling and urine sampling will be performed in enrolled patients prior to implantation of the device(baseline) and at selected follow-ups, to quantify and monitor for systemic Ag release from the prosthetic components. Samples will be appropriately processed and investigated by inductively coupled plasma-mass spectrometry (ICP-MS) analysis.

SECONDARY OUTCOMES:
Clinical scores 1 | day 0 (at baseline), at 1 month follow-up at 3 months follow-up, at 6 months follow-up, at 12 months follow-up, at 24 months follow-up
  The clinical performance of the device through the performance of established clinical scores (Visual analogue scale).
Clinical scores 2 | day 0 (at baseline), at 1 month follow-up at 3 months follow-up, at 6 months follow-up, at 12 months follow-up, at 24 months follow-up
  The clinical performance of the device through the performance of established clinical scores (Short form 36)
Osteointegration | at 1 month follow-up at 3 months follow-up, at 6 months follow-up, at 12 months follow-up, at 24 months follow-up
  The stability and osseointegration of the device through the evaluation of radiological images at different follow-ups (1, 3, 6, 12 and 24 months).
Complications | at 1 month follow-up, at 3 months follow-up, at 6 months follow-up, at 12 months follow-up, at 24 months follow-up
  The occurrence of possible early and late post-implantation complications

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Istituto Ortopedico Rizzoli, Bologna, BO
  - Ospedale Mazzolani Vandini, Argenta, Italia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Akay S, Yaghmur A. Recent Advances in Antibacterial Coatings to Combat Orthopedic Implant-Associated Infections. Molecules. 2024 Mar 6;29(5):1172. doi: 10.3390/molecules29051172. PMID 38474684
- [Background] Chen X, Zhou J, Qian Y, Zhao L. Antibacterial coatings on orthopedic implants. Mater Today Bio. 2023 Feb 15;19:100586. doi: 10.1016/j.mtbio.2023.100586. eCollection 2023 Apr. PMID 36896412
- [Background] Shichman I, Roof M, Askew N, Nherera L, Rozell JC, Seyler TM, Schwarzkopf R. Projections and Epidemiology of Primary Hip and Knee Arthroplasty in Medicare Patients to 2040-2060. JB JS Open Access. 2023 Feb 28;8(1):e22.00112. doi: 10.2106/JBJS.OA.22.00112. eCollection 2023 Jan-Mar. PMID 36864906
- [Background] Tan TL, Maltenfort MG, Chen AF, Shahi A, Higuera CA, Siqueira M, Parvizi J. Development and Evaluation of a Preoperative Risk Calculator for Periprosthetic Joint Infection Following Total Joint Arthroplasty. J Bone Joint Surg Am. 2018 May 2;100(9):777-785. doi: 10.2106/JBJS.16.01435. PMID 29715226
- [Background] Smolle MA, Bergovec M, Scheipl S, Gossler W, Amerstorfer F, Glehr M, Leithner A, Friesenbichler J. Long-term changes in serum silver concentrations after extremity reconstruction with silver-coated megaprostheses. Sci Rep. 2022 Jul 29;12(1):13041. doi: 10.1038/s41598-022-16707-0. PMID 35906279
- [Background] Scoccianti G, Frenos F, Beltrami G, Campanacci DA, Capanna R. Levels of silver ions in body fluids and clinical results in silver-coated megaprostheses after tumour, trauma or failed arthroplasty. Injury. 2016 Oct;47 Suppl 4:S11-S16. doi: 10.1016/j.injury.2016.07.042. Epub 2016 Aug 11. PMID 27523624